CLINICAL TRIAL: NCT02097355
Title: Integrated Clinical Information Sharing System: Implementation and Mixed-Methods Evaluation of a Web-based Monitoring and Management System for Patients With Chronic Conditions
Brief Title: Using an Online Patient Monitoring System to Improve Care for Children With Chronic Conditions
Acronym: TriVoxHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Eugenia Chan, Attending Physician, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: BCH PPQI 52012
Record Dates: First submitted 2014-03-21; First posted 2014-03-27 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Attention Deficit Hyperactivity Disorder; Asthma; Autism Spectrum Disorder; Depression; Epilepsy
Keywords: chronic disease; patient portal; health information technology; patient provider communication; quality improvement
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Asthma; Autism Spectrum Disorder; Depression; Epilepsy; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TriVox Active (Experimental): Provider using TriVox for clinical care
  Interventions: Other: TriVox for clinical care
- TriVox Delayed-start (No Intervention): Providers not using TriVox for clinical care

INTERVENTIONS:
Other: TriVox for clinical care — Use TriVox disease modules to manage patients
  Arms: TriVox Active

SUMMARY:
TriVox Health is an online system designed to make it easy for healthcare providers to monitor patients' disease symptoms and functioning over time and in between in-person visits (http://www.youtube.com/watch?v=VR1vcbx0Ef4). Using combined quality improvement and randomized clinical trial methods, we will evaluate the impact of TriVox on the health outcomes, patient/family experience of care, and healthcare utilization for children and adolescents with Attention Deficit Hyperactivity Disorder (ADHD), asthma, autism, depression, and epilepsy.

DETAILED DESCRIPTION:
TriVox Health is a web-based patient management and monitoring system designed to track patients' disease symptoms and response to therapy over time. TriVox Health enables clinics to use electronic surveys to gather data remotely from multiple responders, including patients, parents/guardians, school personnel and ancillary providers, and view the responses in a timely manner via graphical, tabular, and narrative summary formats.

This quality improvement (QI) initiative will implement TriVox as the standard of care for all patients who receive care for ADHD, asthma, autism, depression, and epilepsy within seven ambulatory specialties at Boston Children's Hospital. Patients and families will use TriVox to report on patient health status and will complete clinically-reTriVoxlevant questionnaires at routine intervals. Providers will use the information collected through TriVox to inform their clinical care of the patient/family.

To evaluate the effectiveness of TriVox, we will conduct a 24-month phased, cluster randomized controlled trial (RCT) where we randomize providers to "active" vs. "delayed-start" to TriVox use, with patients clustered by provider (within specialties) for analytic purposes. Delayed-start providers will crossover to active TriVox use after 12 months. Patients/families will complete additional surveys in order to assess the system's actual or potential effects on patient/family-provider interactions, healthcare utilization and costs.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with clinical diagnosis of ADHD, asthma, autism, depression, and/or epilepsy
* Patient receives care for these diagnoses from providers in participating ambulatory clinics (Primary Care, Adolescent Medicine, Developmental Medicine, Neurology, Psychiatry)
* Patient's primary caregiver enrolled in TriVox

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 946 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in caregiver-rated disease-specific symptoms | Baseline to 12 months
  Caregiver-reported ratings on disease-specific symptom rating scale. For example, Vanderbilt ADHD Parent Rating Scale for ADHD; Asthma Control Test for asthma

SECONDARY OUTCOMES:
Number of patients with "red flag" alerts | 1 month
  Number of patients whose responses to clinical questionnaires trigger a "red flag" alert in ICISS
Change in caregiver-rated global functioning | Baseline to 12 months
  Caregiver ratings on modified Clinical Global Assessment Scale
Experience of care | Baseline and after every ambulatory visit for up to 84 months
  Participant ratings on Post-Visit Experience of Care Survey

OTHER OUTCOMES:
Healthcare utilization | 12 months
  inpatient and ambulatory visits within healthcare system directly related to patient's medical or mental health condition
Direct out of pocket expenditures | 12 months
  Out of pocket expenditures directly related to care for child's medical or mental health condition, e.g. co-pays, prescription costs

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Chan, MD, MPH, Principal Investigator — Boston Children's Hospital; Eric Fleegler, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ICISS: Collaborating Online to Improve Children's Health Care — http://www.youtube.com/watch?v=VR1vcbx0Ef4